CLINICAL TRIAL: NCT00524888
Title: Suturing Vs Adhesion for Hand Lacerations in the ER A Randomized Prospective Study
Brief Title: Suturing vs Biological Adhesive in Simple Lacerations of Hand
Acronym: sutvsglu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sutvsglu-HMO-CTIL
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-08

CONDITIONS: Lacerations
Keywords: Hand; Laceration; bioadhesive; ER; Hand laceration distal to the volar wrist crease
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): suturing lacerations of the hand
  Interventions: Procedure: suturing laceration
- 2 (Active Comparator): using bioadhesive on lacerations of hand
  Interventions: Procedure: bioadhesive

INTERVENTIONS:
Procedure: suturing laceration — suturing simple lacerations of the hand
  Arms: 1
Procedure: bioadhesive — using bioadhesive on simple lacerations of the hand
  Arms: 2

SUMMARY:
To assess the difference in clinical outcome between lacerations in the hand treated by sutures versus treated by tissue adhesive.

ELIGIBILITY:
Inclusion Criteria:

* Any age
* Hand laceration distal to the volar wrist crease.

Exclusion Criteria:

* Fracture , tendon, artery involvement, more than 8 hours from laceration to trx,
* Immunosuppression
* Anticoagulation therapy
* Diabetes
* Unable to achieve homeostasis in more than 15 minutes
* Unwilling to participate in the study
* Unable to participate in the follow up or bite of any kind.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-09

PRIMARY OUTCOMES:
Wound appearance | 3 Months

SECONDARY OUTCOMES:
pain of treatment and time length of treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Icekson, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel